CLINICAL TRIAL: NCT00897559
Title: Identifying the Genetic Basis of Adult AMKL
Brief Title: Study of Bone Marrow Samples From Patients With Acute Leukemia
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000600323; ECOG-E1900T3
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: adult acute megakaryoblastic leukemia (M7)
MeSH Terms: conditions — Leukemia; Leukemia, Megakaryoblastic, Acute | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis; Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymorphism analysis
Genetic: protein analysis
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying the genes expressed in samples of bone marrow from patients with cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking at bone marrow samples from patients with acute leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To perform high throughput sequencing of a set of megakaryocyte specific transcription factors, tyrosine kinases, and Src kinases in DNA isolated from bone marrow specimens of adults with acute megakaryoblastic leukemia (AMKL).
* To assay the ability of Src kinase inhibitors (SU6656, dasatinib) to induce differentiation of AMKL blasts in these patients.

OUTLINE: DNA from previously collected bone marrow samples are sequenced to analyze genes associated with transcription factors (GATA1, GATA2, SCL, FOG-1, ETS1, ETS2, ERG, FLI-1, GABP, HOXA11, NF-E2, and RUNX1), tyrosine kinases (JAK2, JAK3, and c-MPL), and Src family kinases (LYN, FYN, and HCK) and compared with control DNA. Using bioinformatics, gene alterations are compared to known polymorphisms and subsequent changes in the amino acid sequence of the encoded protein. Subsequent assays assess the effect on proliferation and differentiation and in vitro studies evaluate the consequences of mutations on transcription factor and kinase activity abilities. The effect of SU6656 and dasatinib on cell death and polyploidization is evaluated by flow cytometry and compared with control DNA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adult acute megakaryoblastic leukemia
* Archived bone marrow specimens from the ECOG tissue repository

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-07-03; Primary Completion 2009-11-11 (Actual); Study Completion 2009-11-11 (Actual)

PRIMARY OUTCOMES:
Correlation of gene mutations with adult acute megakaryoblastic leukemia (AMKL) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John Crispino, PhD, Study Chair — Robert H. Lurie Cancer Center

IPD SHARING:
Plan to Share IPD: No
Data sharing is dictated by the group's data sharing plan.